## **Pregnancy Partner Informed Consent to Participate in Research**

#### **BMT CTN 1902**

Phase II Multicenter Trial of anti-B Cell Maturation Antigen Chimeric Antigen Receptor T Cell Therapy for Multiple Myeloma Patients with Sub-Optimal Response After Autologous Hematopoietic Cell Transplantation and Maintenance Lenalidomide

| Your Name: | |
|---|---|
| Principal Investigator: | |
| Insert local PI i | nformation |
| Sponsor: | This study is sponsored by the National Institutes of Health, through the Blood and Marrow Transplant Clinical Trials Network |
| The ethics of this | s study have been reviewed and approved by [name of IRB]. |
| ✓ The purp | or or nurse will review this <b>Consent Form</b> with you, including: |
| ✓ The purp | , i |

- ✓ Other options available to you
- ✓ Your rights if you join the study

## 1. Study Overview

You are being asked to provide information on your pregnancy, and on the birth and health of your newborn child, because the biological father of your child is/was participating in a clinical research study titled "Phase II Multicenter Trial of anti-B Cell Maturation Antigen Chimeric Antigen Receptor T Cell Therapy for Multiple Myeloma Patients with Sub-Optimal Response After Autologous Hematopoietic Cell Transplantation and Maintenance Lenalidomide".

The main purpose of this clinical research study is to learn if it is safe and effective (works well) to treat patients who have multiple myeloma with CAR T-cell therapy and maintenance therapy with the drug lenalidomide.

You have become pregnant after the biological father's treatment in this study. The purpose of this consent is to allow collection of information about your pregnancy and newborn by the National Heart, Lung and Blood Institute (NHLBI), who is conducting the research in which your partner participated. Celgene/BMS manufactures the CAR T-cell therapy and information about your pregnancy and newborn will be shared with them. Neither you nor your child will be given any experimental drug if you agree to this consent. We will just collect information from you or your doctor. This information is important to the overall safety evaluation of the CAR T-cell therapy.

If you agree, you may provide this information yourself or give permission to your health care provider and/or obstetrician/gynecologist to release it directly to the biological father's study doctor. If you agree to participate and allow your information to be used and analyzed, you will be asked to sign and date this form.

#### If you agree:

- You or your health care provider will answer questions about your health and your pregnancy.
- We'll collect information through completion of your pregnancy about your health, the pregnancy, and the result of your pregnancy, such as childbirth.
- We'll collect information from your infant's birth through one year of age.

Some possible risks and benefits of joining the study include:

**Possible Risks:** There is a small risk your confidentiality could be lost. The study team will do everything it can to keep your information confidential.

Possible Benefits: None.

If you do **not** join the study, you can continue your usual health care.

### **Key points:**

- Being in any research study is your choice.
- Knowledge gained from this study may help others.
- If you join the study, you can quit at any time. If you decide to quit the study, it will not affect your care at [name of facility or institution].
- Ask the study staff questions about anything you do not understand, or if you would like more information. You can ask questions now or at any time.
- Take time to talk about the study with your doctor, study staff, and your family and friends. It is **your** choice to be in the study. If you decide to join, please sign the end of this Consent Form. You'll get a copy to keep. No one can force you to join this study.

## 2. Study Purpose

We are completing the study the biological father is/was a part of to see if CAR T-cell therapy and maintenance therapy with the drug lenalidomide can help delay multiple myeloma from coming back.

**CAR T-cell therapy** is a treatment made of the biological father's own immune cells (or T cells). CARs, or chimeric antigen receptors, are added to the T cells in a lab. Doctors think that these receptors will help the biological father's T-cells find and attack the myeloma cells.

The specific CAR T-cell therapy in this study, bb2121, has **not** been approved by the U.S. Food and Drug Administration (FDA) to treat multiple myeloma that has already been treated. This study is registered with the FDA, and they will monitor it for safety.

The purpose of this consent is to learn if exposure to CAR T-cell therapy affects an unborn baby. The biological father has received CAR T-cell therapy. At this time, it is not known whether CAR T-cell therapy has an effect on an unborn baby or sperm. The biological father may have also received lenalidomide. Lenalidomide can cause severe birth defects or death of a baby if the father is taking this medicine at the time of conception.

## 3. Study Treatment and Tests

The biological father's study doctor will **not** do any examinations, tests, or procedures on you.

You or your health care provider will answer questions about you and your pregnancy, and we

will collect information from your medical records.

We will collect information about:

- Your age, sex, and race/ethnicity
- Your physical or mental health
- Any medicines that you take during your pregnancy
- Any previous pregnancies, including any complications
- Your current pregnancy
- Your delivery
- Your baby's health

If you have an abortion or a miscarriage, we'll ask for health information from you or your doctor so we can learn if the study treatment affects pregnancy.

#### 4. Risks and Benefits

## **Possible Benefits**

You will receive no benefits or payment for joining this study. The information we learn may help us care for people in the future who become pregnant after they or their partner has received CAR T-cell therapy or lenalidomide.

#### **Possible Risks**

There are very few risks with sharing your medical information and answering questions about your pregnancy. The main risk is that your confidentiality could be lost. The study team will do everything it can to keep your answers confidential.

## 5. Your Rights to Withdraw, Ask Questions, and Seek Other Treatment

Agreeing to provide information about your pregnancy and newborn is your choice. You can choose **not** to provide medical information. If you initially agree to provide information you can change your mind at any time. If you choose to not participate, it won't affect your regular medical care in any way. If at any time you are considering leaving the study, talk to your study doctor about your health and safety.

If you do **not** want to share information about your pregnancy, you may still contact the study doctor at any time to get updated information about the safety of CAR T-cell therapy and lenalidomide.

You have the right to ask questions about the study at any time. If you have questions about the study, please contact:

## [Insert contact details of Principal Investigator or Study Team]

If you want to talk with someone not directly involved in the study, or have any complaints or questions about your rights as a research participant or about potential risks and injuries, you may contact the NMDP IRB Administrator at:

1-800-526-7809

You must tell [insert name of Principal Investigator] if you decide to leave the study.

## **6.** New Information Available During the Study

During the study the biological father is/was a part of, the study doctors may learn new information about CAR T-cell therapy and the risks to pregnancy or babies. If they learn new information, they'll tell you or the biological father as soon as it's available.

## 7. Privacy, Confidentiality, and Use of Information

Your privacy is very important to us. The study doctors, study sponsor, and other groups with access to your pregnancy-related medical information will do everything they can to protect it. The study doctors can protect your records if there is a court case. However, some of your medical information may be shared if required by law. If this happens, the study doctors will do their best to make sure that any information that goes out to others will **not** identify you or your newborn.

Your confidentiality is one of our main concerns. We will do our best to make sure that the personal information in your medical record is kept confidential (private). However, we cannot promise total privacy.

To make sure the study is running ethically, some government agencies or other groups may need to access part of your medical records. For this study, those groups include:

#### [Institution]

- The National Institutes of Health (NIH), which include the National Heart, Lung, and Blood Institute (NHLBI) and the National Cancer Institute (NCI)
- U.S. government agencies that are responsible for overseeing research such as the Food and Drug Administration (FDA) and the Office of Human Research Protection (OHRP)
- U.S. government agencies that are responsible for overseeing public health concerns such as the Centers for Disease Control (CDC) and federal, state, and local health departments

- The Data and Safety Monitoring Board (DSMB), not part of [Institution]
- The National Marrow Donor Program (NMDP) Institutional Review Board (IRB) responsible for this study
- Blood and Marrow Transplant Clinical Trials Network (BMT CTN) Data and Coordinating Center (DCC), including:
  - The Center for International Blood and Marrow Transplant Research (CIBMTR)
  - The NMDP
  - Emmes, a company that coordinates the BMT CTN studies
- Celgene/BMS, its collaborators, or designees. This may include people within or outside of the United States (U.S.). Privacy laws outside of the U.S. may be less strict.
- Study investigators

If information regarding pregnancy from the biological father's study is published or presented at scientific meetings, your name and other personal information will not be used. Study information may also be used for research in the future.

A description of the biological father's clinical study is available on <a href="http://www.clinicaltrials.gov">http://www.clinicaltrials.gov</a>. This website does not include information that can identify the biological father or you. You can search this website at any time.

## 8. Leaving the Study

You may choose to no longer provide pregnancy or newborn information at any time.

If you leave, the information already collected from you will still be included in the biological father's study. If you don't want your information to be used, you **must** let his study doctor know.

#### 9. Cost and Reimbursement

You will receive **no** benefits or payment for providing information to the biological father's study. This research will not cover any costs related to your pregnancy, delivery, newborn care, abortion, or miscarriage.

# 10. Health Insurance Portability and Accountability Act 1 (HIPAA) Authorization to use health information for research

Your local study site will give you a separate form with information about the Health Insurance

Portability and Accountability Act 1 (HIPAA).

**TITLE**: BMT CTN 1902: Phase II Multicenter Trial of anti-B Cell Maturation Antigen Chimeric Antigen Receptor T Cell Therapy for Multiple Myeloma Patients with Sub-Optimal Response After Autologous Hematopoietic Cell Transplantation and Maintenance Lenalidomide

- I have read and understood this Consent Form. The purpose and description of the information requested has been explained to me.
- I have had the chance to ask questions and understand the answers I have been given. I understand that I may ask questions at any time.
- I freely agree to provide pregnancy information to my partner's study.
- I have had the chance to discuss my participation with a family member or friend if I choose.
- I understand that...
  - o I may not directly benefit from providing pregnancy or newborn medical information.
  - My name and personal information will not be identified even if information gained is published.
  - o I can stop providing medical information at any time and doing so will not affect my current care or prevent me from receiving future treatment.
  - o I will be given a copy of this signed consent form.
  - o I do not give up any legal rights by signing this form.

| Participant Name (or Parent/Guardian) | Date (MM/DD/YYYY) |
|--------------------------------------------|-------------------|
| Participant Signature (or Parent/Guardian) | Date (MM/DD/YYYY) |

## Physician certification

| I certify that I have provided a verbal explanation of the determinant the procedures and risks. I believe the participant has under | · · |
|---|---|
| Counseling Physician Name | Date (MM/DD/YYYY) |
| Counseling Physician Signature | Date (MM/DD/YYYY) |
| Interpreter certification (if needed) I certify that I have provided an accurate interpretation of participant has understood the information provided. | this consent form. I believe the |
| Interpreter Name | Date (MM/DD/YYYY) |
| Interpreter Signature | Date (MM/DD/YYYY) |